CLINICAL TRIAL: NCT05100979
Title: Patient-Clinician Communication Skill Training: A Mobile Education Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mir A Basir, Professor of Pediatrics, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00040976
Record Dates: First submitted 2021-10-07; First posted 2021-10-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Communication; Patient Engagement
Keywords: mobile health; medical education; patient-clinician communication
MeSH Terms: conditions — Communication; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art of Medicine Series (Experimental): Participants receiving the Art of Medicine Series will be sent text messages throughout the 4 week study intervention period. Each text message contains a link to a short, animated video teaching an evidence-based communication technique.
  Interventions: Other: The Art of Medicine Series

INTERVENTIONS:
Other: The Art of Medicine Series — The Art of Medicine Series is a smartphone-based educational tool focused on teaching communication strategies to clinicians and patients.

SUMMARY:
This study is a pilot test of The Art of Medicine Series, a smartphone-based educational tool to improve clinician-patient communication. Investigators will enroll clinicians (residents, fellows, attending physicians) and family caregivers (most often parents) from the Children's Wisconsin neonatal intensive care unit (NICU). Participants will then receive a series of links to short, animated videos sent to their phone by text message. Each video teaches best-practice communication techniques such as how patients can prompt teach back and how clinicians can avoid biased phrasing in delivering news. Over the 4-week intervention (the length of resident's rotation), clinicians will receive 15 videos and patients will receive 8 videos. Communication skills of clinicians and patients will be assessed pre and post intervention using validated measures and participants' engagement with the videos will be tracked with software in the website.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria - clinician:

* A resident, fellow, or attending physician
* On Team A rotation in the neonatal intensive care unit (NICU) of Children's Wisconsin.

Inclusion criteria - patient:

* A parent, grandparent, or other identified caregiver of a child on Team A of the NICU at Children's Wisconsin
* Expected to stay in the NICU for a further 3 weeks
* Have not previously participated in the study
* Are 18 years of age or older
* Able to speak and understand English.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Clinician communication skills | Assessed at 4 weeks
  Clinician communication skills are primarily measured using the validated Gap Kalamazoo Communication Skills Self-Assessment.
Patient communication skills | Assessed at 4 weeks
  Patient (family caregiver) communication skills are primarily measured using the • Perceived Self-Efficacy in Patient-Physician Interactions (PEPPI).

SECONDARY OUTCOMES:
Participant engagement with videos | Collected at 4 weeks
  Participant (both clinician and patient) engagement with videos is measured through tracking software on The Art of Medicine Series website.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No